CLINICAL TRIAL: NCT04355416
Title: Clinical Evaluation of 1% Curcumin Oral Gel and Its Effect on the Clinical Attachment Level and the Level of IL-8 in GCF in Treatment of Periodontal Pocket
Brief Title: Clinical and Anti-inflammatory Effect of Curcumin Oral Gel as Adjuncts in Treatment of Periodontal Pocket
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Baghdad (Other)
Collaborators: Najaf dental specialized center (Unknown)
Responsible Party: Principal Investigator, Haider Thabit, Specialist dentist, University of Baghdad
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Health Services Research
Other Study IDs: college of dentistry
Record Dates: First submitted 2020-04-15; First posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Chronic Periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Dental Scaling; Root Planing

STUDY DESIGN:
Intervention Model Description: Twenty five systemically healthy patients either male or female with chronic periodontitis aged between 30 and 45 years with pocket depth of 5-7 mm affecting at least two nonadjacent sites will be included. A split mouth design will be followed Selected sites will be randomized into control and experimental sites. In the experimental site scaling and root planing to be performed, followed by placement of the curcumin gel and periodontal pack application. In the control site, sub gingival scaling and root planing alone will be performed followed by periodontal pack application. collecting of GCF from the pocket to determine the level of IL_8 by ELISA and measurement of the clinical Parameters to be included: PLI (plaque index), BOP (bleeding on probing), PPD (probing pocket depth) and RAL (relative attachment level). These parameters will be recorded on day 0 and 30 days.
Who Masked: Care Provider
Masking Description: care provider not involved in the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- curcumin oral gel (Experimental)
  Interventions: Drug: curcumin Oral gel; Procedure: subgingival scaling and root planing
- subgingival scaling and root planing (Other)
  Interventions: Procedure: subgingival scaling and root planing

INTERVENTIONS:
Drug: curcumin Oral gel — application of curcumin oral gel after scaling and root planing
  Arms: curcumin oral gel
Procedure: subgingival scaling and root planing — subgingival scaling and root planing without application of curcumin gel

SUMMARY:
application of 1% curcumin gel in clinical study design will be used . The study will be conducted in Al-Najaf specialised dentistry center. The group of patients will be consist of 25 patients, belonging to both sex, age between 30-45 years. All patients will be diagnosed as chronic periodontitis with periodontal pockets of depth 5-7mm bilaterally to be randomly selected.

DETAILED DESCRIPTION:
Abstract:

Background: Complete removal of irritants is not possible with mechanical therapy alone. Adjunctive use of systemic administration of antibiotics results in the distribution of drug throughout the body, which can give rise to toxicity. Curcumin (diferuloylmethane), a constituent of Curcuma longa plant, which possess antioxidant, anti-inflammatory, and anti-microbial properties. The aim of the study is to determine the effect of curcumin oral gel on the anti-inflammatory chemokines (IL_8) in the gingival crevicular fluid and to compare the effects of the curcumin gel as an adjunct to sub gingival scaling and root planing with the effect achieved using sub gingival scaling and root planing alone.

Twenty systemically healthy patients either male or female with chronic periodontitis aged between 30 and 45 years with pocket depth of 5-7 mm affecting at least two nonadjacent sites will be included. A split mouth design will be followed and the patients will receive a complete prophylaxis including scaling and root planning. In the experimental site scaling and root planing to be performed, followed by placement of the curcumin gel and periodontal pack application. In the control site, sub gingival scaling and root planning alone will be performed followed by periodontal pack application. collecting of GCF from the pocket which will be followed the same site for each visit to determine the level of IL_8 by ELISA and measurement of the clinical Parameters to be included: PLI (plaque index), BOP (bleeding on probing), PPD (probing pocket depth) and RAL (relative attachment level). These parameters will be recorded on day 0 and 30 days.

The aim of the study :

To determine the effect of curcumin oral gel on the anti inflammatory chemokines (IL_8) in the gingival crevicular fluid and to compare the effects of the curcumin gel as an adjunct to sub gingival scaling and root planning with the effect achieved using sub gingival scaling and root planing alone in the treatment of (5-7 mm) periodontal pockets on clinical Parameters: PLI (plaque index), BOP (bleeding on probing) , PPD (probing pocket depth) and RAL (relative attachment level).

Objectives:

1. To evaluate the efficacy of sub gingival application of curcumin gel as an adjunct to SRP in the treatment of (5-7 mm) periodontal pockets on clinical periodontal parameter.
2. To measure the concentration of IL-8 in gingival crevicular fluid before and after treatment.

Hypothesis:

Curcumin gel may have anti-inflammatory effect by reducing IL-8 and may have effect on clinical Parameters: PLI (plaque index), BOP (bleeding on probing) , PPD (probing pocket depth) and RAL (relative attachment level) in the treatment of periodontal pockets .

Alternative hypothesis:

There may be no difference in treatment of periodontal pocket by scaling and root planning and by scaling and root planning adjunct by curcumin oral gel.

Methodology:

Study design: Double blind, prospective , bio clinical research.

Setting: AL-Najaf dental specialized center.

Study design and population:

Twenty systemically healthy patients either male or female with chronic periodontitis aged between 30 and 45 years with pocket depth of 5-7 mm affecting at least two nonadjacent sites will be included. A split mouth design will be followed and the patients will receive a complete prophylaxis including scaling and root planing. Selected sites will be randomized into control and experimental sites. In the experimental site scaling and root planing to be performed, followed by placement of the curcumin gel and periodontal pack application. In the control site, sub gingival scaling and root planing alone will be performed followed by periodontal pack application. collecting of GCF from the pocket which will be followed the same site for each visit to determine the level of IL_8 by ELISA and measurement of the clinical Parameters to be included: PLI (plaque index), BOP (bleeding on probing), PPD (probing pocket depth) and RAL (relative attachment level). These parameters will be recorded on day 0 and 30 days.

Procedure/intervention:

collecting of GCF from the pocket which will be followed the same site for each visit to determine the level of IL_8 by ELISA and measuring of the clinical parameters: PLI (plaque index), BOP (bleeding on probing) , PPD (probing pocket depth) and RAL (relative attachment level) prior to the each procedure. The pocket will randomly have selected for both groups. PD will be measured with UNC 15 mm probe, acrylic stent as a guide for reproducibility from the gingival margin to base of the pocket. To achieve concealment, the patient will be blinded about intervention which side is test and which side is control. Before baseline (baseline regarded as first visit) we do oral hygiene motivation and supra gingival scaling only. At first visit (baseline ) day 0 will include collecting GCF from pocket of both side ( test and control ) to determine the level of IL_8 by ELISA and measurement of the clinical parameters : PLI (plaque index) , BOP (bleeding on probing), PPD (probing pocket depth) and RAL (relative attachment level) it also include sub gingival scaling and root planing for both side and curcumin gel will be inserted to the pocket of tested group with a 2 ml disposable syringe equipped with a blunted 25-gauge needle, which is bent along its shank after that periodontal dressing (Coe- Pak) will be used to cover the pocket on both side so as to prevent the ingress of oral fluids as well as to allow the retention of the material within the pocket. The first visit will also include oral hygiene instructions. Subjects will be recalled after 7 days, for periodontal dressing to be removed and curcumin gel will be inserted to the pocket of tested group.

The second visit (after thirty day)will include collecting GCF from the same previous site of pocket on both side to determine the level of IL_8 by ELISA and measurement of the clinical parameters : PLI (plaque index) , BOP (bleeding on probing), PPD (probing pocket depth) and RAL (relative attachment level).To ensure excellent collection of GCF, we must make sure the sites should be dried and not contaminated by saliva or blood, using cotton rolls, gentle force should be applied to avoid bleeding and the periocol strip should be inserted for 30 seconds, the sample will be transferred into eppendrof tubes and stored in -20 c until the completion of the samples collections, the tube will be allocated to the patient'code.

Assessment of the clinical parameters in the recall visit, separation of the GCF will be done by the following procedure : each sample will be micro centerfuged at 400-500g for 4-5 min then diluted by 500 microliter phosphate buffered saline and stored overnight in 4c to achieve optimal protein elusion. the periocol is then removed and the supernatants will be assayed by ELISA.

The total level of the IL_8 will be determined by using ELISA kits according to the manufacture instruction.

ELIGIBILITY:
Inclusion Criteria:

1. Age group of 30-45 years.
2. Belonging to both sexes.
3. Chronic periodontitis patients.
4. Probing pocket depth (PPD) 5-7 mm.

Exclusion Criteria:

1. Subjects having taken antibiotics prior to or during the trial.
2. Patients on medication likely to induce gingival enlargement.
3. Pregnant or lactating women.
4. Smokers.
5. Tobacco chewers.
6. Allergy to curcumin oral gel.
7. Patients with systemic disease.

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2020-04-20 (Actual); Primary Completion 2020-05-30 (Estimated); Study Completion 2020-06-30 (Estimated)

PRIMARY OUTCOMES:
measuring interleukin -8 | one month
  measuring interleukin -8 in gingival crevicular fluid by using ELISA
measuring plaque accumulation | one month
  measuring plaque accumulation on the teeth by measuring the plaque index using periodontal probe
measuring gingival inflammation | one month
  measuring gingival inflammation by measuring the gingival index by using periodontal probe
measuring periodontal pocket erosion | one month
  measuring periodontal pocket erosion and destruction by measuring bleeding on probing index using periodontal probe
measuring the periodontal pocket depth | one month
  measuring the periodontal pocket depth by using periodontal pocket depth index using periodontal probe
measuring periodontal attachment level | one month
  measuring periodontal attachment level by measuring clinical attachment level index using periodontal probe

CONTACTS AND LOCATIONS:
Locations (1):
- university of Baghdad college of dentistry, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: Undecided